CLINICAL TRIAL: NCT05986604
Title: NIA_Improving Sleep and Circadian Functioning, Daytime Functioning, and Well-being for Midlife and Older Adults by Improving Patient Memory for a Transdiagnostic Sleep and Circadian Treatment
Brief Title: NIA_Improving Function and Well-being by Improving Patient Memory: Transdiagnostic Sleep and Circadian Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TranS-C+MSI vs. TranS-C Alone
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disorder; Circadian Dysregulation; Memory Impairment
MeSH Terms: conditions — Sleep Wake Disorders; Chronobiology Disorders; Memory Disorders | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to TranS-C plus the MSI ("TranS-C+MSI") or TranS-C alone
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TranS-C+MSI (Experimental): Transdiagnostic Intervention for Sleep and Circadian Dysfunction will be combined with the Memory Support Intervention
  Interventions: Behavioral: Memory Support Intervention; Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction
- TranS-C alone (Active Comparator): The Transdiagnostic Sleep and Circadian Intervention will be delivered alone
  Interventions: Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction

INTERVENTIONS:
Behavioral: Memory Support Intervention — The Memory Support Intervention is designed to improve patient memory for treatment and involves a series of specific procedures that support the encoding and retrieval stages of episodic memory. The memory support strategies are proactively, strategically and intensively integrated into treatment-as-usual to support encoding. Memory support is delivered alongside each 'treatment point', defined as a main idea, principle, or experience that the treatment provider wants the patient to remember or implement as part of the treatment.
  Other Names: MSI
  Arms: TranS-C+MSI
Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction — TranS-C aims to provide one protocol to treat a range of sleep and circadian problems because sleep and circadian problems are often not so neatly categorized and because the existing research provides few guidelines to treat more complex patients.
  Other Names: TranS-C

SUMMARY:
Mental illness is often chronic, severe, and difficult to treat. Though there has been significant progress towards establishing effective and efficient interventions for psychological health problems, many individuals do not gain lasting benefits from these treatments. The Memory Support Intervention (MSI) was developed utilizing existing findings from the cognitive science literature to improve treatment outcomes. In this study, the investigators aim to conduct an open trial that includes individuals 50 years and older to assess if a novel version of the Memory Support Intervention improves sleep and circadian functioning, reduces functional impairment, and improves patient memory for treatment.

DETAILED DESCRIPTION:
Life expectancy has increased drastically in the United States. Longer life is too often associated with illness, discomfort, disability, and dependency. Progress toward promoting health and well-being as we age must include the identification of novel treatment targets that are safe, powerful, inexpensive, and deployable. The proposed research will test one such target-patient memory for the contents of treatment.

Over 5 years, we will recruit adults who are 50 years and older and who are experiencing sleep and circadian problems (n = 178, including 20% for attrition). Participants will be randomly allocated to TranS-C plus the MSI ("TranS-C+MSI") or TranS-C alone via eight 50-minute, weekly, individual sessions. Assessments will be conducted at baseline, post-treatment, and at 6- and 12-month follow-up (6FU and 12FU).

Specific Aim 1: To evaluate if adding the MSI to TranS-C (a) improves sleep and circadian functioning, (b) improves daytime functioning, (c) improves well-being and (d) improves patient memory by comparing the effects of TranS-C+MSI vs. TranS-C alone. Hypothesis 1. Compared to TranS-C alone, people who receive TranS-C+MSI will improve more on all outcomes at post-treatment, 6FU and 12FU.

Specific Aim 2: To evaluate if patient memory for treatment mediates the relation between treatment condition and sleep and circadian functioning. Hypothesis 2. TranS-C+MSI will be associated with better memory for treatment relative to TranS-C alone, and in turn, better memory for treatment will be associated with better sleep and circadian functioning immediately following treatment and at 6FU and 12FU.

Specific Aim 3: To evaluate if subgroups hypothesized to derive added benefit from memory support moderate (a) patient memory for treatment and (b) treatment outcome. Hypothesis 3. Treatment effects for TranS-C+MSI will be larger at post-treatment for those who are older, have fewer years of education, poorer baseline cognitive functioning and more severe baseline sleep disruption and sleep-related impairment.

Exploratory analyses will compare the treatments on (a) patient adherence as well as patient-rated treatment credibility and utilization of treatment elements and (b) provider-rated acceptability, appropriateness, and feasibility.

ELIGIBILITY:
Inclusion criteria:

1. Aged 50 years and older;
2. English language fluency;
3. Experiencing a mobility impairment;
4. Low income;
5. Exhibit a sleep or circadian disturbance as determined by endorsing 4 "quite a bit" or 5 "very much" (or the equivalent for reverse scored items) on one or more PROMIS-SD questions.
6. 25-30 on the Montreal Cognitive Assessment, as a negative screen for cognitive impairment.
7. Able/willing to give informed consent.

Exclusion criteria:

1. Severe untreated sleep disordered breathing (AHI>30) or moderate untreated sleep disordered breathing with severe daytime sleepiness (AHI of 15-30 and Epworth Sleepiness Scale >10);
2. Medical conditions that prevent a participant from comprehending and following the basic tenants of treatment (e.g., dementia) or that interfere with sleep in a manner that can't be addressed by a cognitive behavioral treatment (e.g., the Structured Clinical Interview for Sleep Disorders will be used to screen for narcolepsy, REM sleep behavior disorder) or that may preclude full participation (e.g., receipt of end of life care);
3. Homelessness;
4. Night shift work >2 nights per week in the past 3 months;
5. Substance abuse/dependence only if it makes participation in the study unfeasible;
6. Suicide risk sufficient to preclude treatment on an outpatient basis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-07-28 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Sleep Disturbance | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Assesses perceived functional impairments related to sleep problems using a self-report questionnaire. The minimum value is 8. The maximum value is 40. Higher scores mean more sleep disturbance (worse outcome).
Sheehan Disability Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Assesses functional impairment on a scale from 0 to 30, where higher scores mean higher impairment
Satisfaction with Life Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  5-item instrument designed to measure global cognitive judgements of satisfaction with one's life. Scores can range from 5-35 with higher scores indicating higher levels of satisfaction with life.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Assesses perceived functional impairments related to sleep problems in a self-report questionnaire. The minimum value is 16. The maximum value is 80. Higher scores mean more sleep related problems (worse outcome).
Positive and Negative Affect Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Positive affect scores can range from 10-15, with higher scores representing higher levels of positive affect. Negative affect scores can range from 10-50, with lower scores representing lower levels of negative affect
WHODAS 2.0 | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  A measure of functional impairment
Cognitive Failures Questionnaire | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Used to assess the frequency with which people experienced cognitive failures. Scores range from 0-100, with higher scores indicating higher levels of cognitive failures.
Epworth Sleepiness Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Used to assess daytime sleepiness. Scores can range from 0-24 with higher scores indicating higher levels of daytime sleepiness.
Memory for Treatment: Cumulative recall | Week 4 of treatment as well as Post Treatment, defined as two weeks after the final therapy session (i.e. 8-10 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up]
  Recall on the Patient Treatment Recall Task
Thoughts and Applications Task | Week 4 of treatment as well as Post Treatment, defined as two weeks after the final therapy session (i.e. 8-10 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up]
  Measures how treatment points have generalized to the participant's thinking and functioning during every day life
Adapted Utilization Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  19-item; 0-4 scale. Scores can range from 0 to 76 (Higher score means more utilization).
Composite Sleep Health Score | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Composite Sleep Health Score which is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint fluctuation), Satisfaction (Sleep quality question on PROMIS-SD), Alertness (Daytime sleepiness question on PROMIS-SRI), Timing (Mean midpoint), Efficiency (Sleep efficiency) and Duration (Total Sleep Time).
Mean sleep efficiency (Daily Sleep Diary) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Daily Sleep Diary mean for sleep efficiency (total sleep time/time in bed X 100)
Mean total wake time (Daily Sleep Diary) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Daily Sleep Diary mean for total wake time defined as sleep onset latency + wake after sleep onset + Early morning awakening
Mean for total sleep time (Daily Sleep Diary) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment to 6-month follow-up to 12-month follow-up
  Daily Sleep Diary mean for total sleep time
Mean for total wake time (Actigraphy) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Actigraphy mean for total wake time defined as sleep onset latency + wake after sleep onset + early morning awakening
Mean for total sleep time (Actigraphy) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Actigraphy mean for total sleep time
Mean for daytime activity (Actigraphy) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Actigraphy mean for daytime activity
Provider level: Acceptability of Intervention Measure | Through therapy completion, an average of 8 weeks following baseline
  Assess provider perceptions of the acceptability of the treatment intervention using a self-report questionnaire
Provider level: Appropriateness Intervention Measure | Through therapy completion, an average of 8 weeks following baseline
  Assesses provider perceptions of the appropriateness of the treatment intervention using a self-report questionnaire
Provider level: Feasibility of Intervention Measure | Through therapy completion, an average of 8 weeks following baseline
  Assesses provider perceptions of the feasibility of the intervention using a self-report questionnaire
Provider level: Provider-rated TranS-C Checklist | Every treatment session which is 8 sessions, spaced one week apart for approximately 8-10 weeks
  A measure of the TranS-C elements that are delivered. This is completed by the therapist at the end of every treatment session
Provider level: Memory Support Treatment Provider Checklist | Every treatment session which is 8 sessions, spaced one week apart for approximately 8-10 weeks
  A measure of memory support delivered. This is completed by the therapist at the end of every treatment session
Provider level: Patient adherence via the TARS | Every treatment session which is 8 sessions, spaced one week apart for approximately 8-10 weeks
  A measure of patient treatment adherence completed by the therapist at the end of every treatment session
Provider level: Memory Support Rating Scale, total amount | Randomly selected therapy tapes
  Assesses the total amount of memory support used by a provider via coding of session tapes
Provider level: Memory Support Rating Scale, number of types | Randomly selected therapy tapes
  Assesses the number of types of memory support used by a provider via coding of session tapes

OTHER OUTCOMES:
WatchPAT One | Baseline only
  For participants who screen positive for obstructive sleep apnea, WatchPAT One will be offered to determine eligibility
Adverse events checklist | Only at post-treatment which is 8-10 weeks after the beginning of treatment
  To assess any adverse events experienced as a result of participating in the study
Montreal Cognitive Assessment (MoCA) | Baseline only
  A measure of cognitive functioning/cognitive impairments to determine eligibility
Adapted Credibility Expectancy Questionnaire | At treatment Week 2 and at post-treatment which is 8-10 weeks after the beginning of treatment
  Measures the credibility and expectation of improvement from the treatment.
Structured Clinical Interview for Sleep Disorders | Baseline only
  Measures sleep and circadian diagnoses according to DSM-5
Adapted Brief Disability Questionnaire | Baseline only
  A measure of functional impairment

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Milner AE, Hache RE, Oliver S, Sarfan LD, Spencer JM, Cogan A, Jiang Y, Agnew ER, Zieve GG, Martin JL, Zeidler MR, Dong L, Carpenter JK, Varghese J, Bol K, Bajwa Z, Tighe CA, Harvey AG. Integrating the Memory Support Intervention into the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): can improving memory for treatment in midlife and older adults improve patient outcomes? Study protocol for a randomized controlled trial. Trials. 2024 Oct 3;25(1):650. doi: 10.1186/s13063-024-08468-0. PMID 39363383